CLINICAL TRIAL: NCT00860392
Title: A Comparison of Measurements of Ketone Body Flux Versus Ketone Body Concentration as a Pharmacodynamic Marker of Hepatic Fatty Acid Oxidation
Brief Title: A Comparison of Measurements of Ketone Body Flux Versus Ketone Body Concentration as a Pharmacodynamic Marker of Hepatic Fatty Acid Oxidation (0000-110)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-110; 2009_560
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Biomarker evaluation
  Interventions: Drug: Stable isotope tracer (13-C(4)-BHB)

INTERVENTIONS:
Drug: Stable isotope tracer (13-C(4)-BHB) — A stable isotope tracer (13-C(4)-BHB), a commercially available lipid emulsion, and heparin will be administered intravenously. Ketone body concentrations will be measured before beginning the infusion, at approx. 135 minutes, and at approx. 255 minutes.

SUMMARY:
This study will compare two approaches to the measurement of fatty acid oxidation (ketone body flux and ketone body concentration) and determine which method demonstrates superior sensitivity and variability in the detection of moderate increases in ketogenesis rates.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index of 18-25 kg/m2 OR 29-40 kg/m2
* Subject has been a nonsmoker or has not used nicotine for the past 6 months

Exclusion Criteria:

* Subject has a history of diabetes mellitus
* Subject has a history of stroke, chronic seizures, or other neurological disorder
* Subject has a history of cancer, except certain skin cancers
* Subject consumes more than 3 alcoholic beverages per day
* Subject consumes more than 6 servings of caffeinated beverages per day
* Subject has multiple and/or severe allergies to food or drugs
* Subject has allergy or sensitivity to eggs or soy
* Subject regularly uses illicit drugs or has a history of drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2009-07-08 (Actual); Study Completion 2009-07-08 (Actual)

PRIMARY OUTCOMES:
Effects of increase in serum free fatty acid levels on ketogenesis as measured using a isotopic tracer and serum ketone body concentration in healthy lean subjects | 5 hours

SECONDARY OUTCOMES:
Effects of increase in serum free fatty acid levels on ketogenesis as measured using a isotopic tracer and serum ketone body concentration in obese subjects | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC